CLINICAL TRIAL: NCT01012648
Title: Early Fluid Resuscitation With Balanced HES 130/0.4 [6%] in Severe Burn Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Béchir Markus, MD, Intensivmedizin
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BURN
Record Dates: First submitted 2009-10-29; First posted 2009-11-13 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Fluid resuscitation — Volume resuscitation
Drug: HES 130/0.4 (6%), Voluven balanced vs. Lactated Ringer's solution — Volume Resuscitation

SUMMARY:
RCT colloids versus cristalloids only in severe burn victims.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Deep burn injury more than 15% of total body surface area (2nd and 3rd degree burns)
* Informed consent (via deferred consent, if necessary, according to Swiss HMG § 55 and 56).
* Patients or relatives can understand the study information and the provided information in German language

Exclusion criteria:

* Patients expected to succumb within the next 24 to 36 hours, i.e. whole body burn trauma, palliative care situation
* Pregnancy
* No informed consent
* Known allergic reaction to HES
* Patients or patient's relatives, who do not understand the German language and therefore the study information, can not be provided in a legally correct manner.
* Patients with contraindications for balanced 6% HES 130/0.4, i.e. heart failure, pulmonary edema, intracerebral bleeding, acute renal failure, severe hypernatraemia and other severe electrolyte imbalances, severe von-Willebrand Syndrome and acute liver failure (see "Arzneimittelkompendium der Schweiz® - Documed")

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Reduced amount of fluids given | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Markus Béchir, M.D:, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- Surgical ICU, Zurich, Switzerland

REFERENCES:
- [Derived] Bechir M, Puhan MA, Fasshauer M, Schuepbach RA, Stocker R, Neff TA. Early fluid resuscitation with hydroxyethyl starch 130/0.4 (6%) in severe burn injury: a randomized, controlled, double-blind clinical trial. Crit Care. 2013 Dec 23;17(6):R299. doi: 10.1186/cc13168. PMID 24365167